CLINICAL TRIAL: NCT06047652
Title: Electronic Continuing Professional Development (e-CPD) Implementation, Process, and Outcomes for Indonesian Clinical Nurses: An Exploratory Action Research Study Protocol.
Brief Title: Development of Electronic Continuing Professional Development for Indonesian Clinical Nurses
Acronym: e-CPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitas Muhammadiyah Yogyakarta (Other)
Responsible Party: Principal Investigator, Novita Kurnia Sari, Assistant Professor, Universitas Muhammadiyah Yogyakarta
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: e-CPD dev
Record Dates: First submitted 2023-08-25; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Nurse's Role
Keywords: exploratory action research; electronic learning; continuing professional development; protocol; nurse

STUDY DESIGN:
Intervention Model Description: This study is a seven-stage exploratory action research, with stage 6 being the Moodle e-CPD trial for hospital nurses.
Masking Description: This study consists of 4 participant groups, of which 3 will conduct FGDs to investigate data and 1 will conduct Moodle e-CPD trials. The four categories of participants are nurses with experience implementing CPD, hospital management responsible for implementing CPD for nurses, members of the Indonesian nursing professional organization with the authority to manage CPD for nurses, and clinical nurses with at least level 1 certification. However, the Moodle e-CPD trial will only be conducted with a group of at least level 1 clinical nurse participants.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): The e-CPD device will be given to the participant group according to the criteria. Each participant is given access rights for 1 week to try all the features in e-CPD.
  Interventions: Device: e-CPD user testing

INTERVENTIONS:
Device: e-CPD user testing — nurses who meet the criteria will carry out user testing on the e-CPD application via a mobile device. after accessing the e-CPD system the nurse will fill in the System Usability Scale instrument.

SUMMARY:
The goal of this clinical trial is to test a e-CPD prototype device for feasibility as it is applied within the clinical nursing setting in Level II clinical nurses in Indonesia. The main questions it aims to answer are:

* What are the user needs for clinical nurse e-CDP development?
* How is an instructional design developed for the development of e-CPD for clinical nurses?
* What is the most suitable e-CPD format for clinical nurses?
* How is the feasibility of e-CPD prototype?

DETAILED DESCRIPTION:
This research is an exploratory action research. This design is principally exploratory research (plan to explore - explore - analyse, and reflect) followed by action research (plan to change - act - observe - reflect)

1. Exploration

   This stage includes the plan to explore stage or stage 1 of 7 research stages. This stage prepares before collecting data. Researchers will start by building good interpersonal relationships with participants and the research environment. A good relationship can also create trust to improve the quality of the data collected. At this stage, researchers also compiled interview guidelines for 3 groups of participants.

   The next stage is exploring, which is stage 2 of the 7 stages of existing research. This stage conducts data collection through FGD to 3 groups of participants. The explanation of the implementation of the FGD is as follows:

   FGD on nurses will be conducted on 8-10 nurses who have performed CPD and have followed the credentials carried out by the hospital. The purpose of this FGD with nurses is to explore understanding, experience, obstacles, efforts made to overcome obstacles, and expectations on the implementation of CPD.

   FGD on hospital management will be conducted on 8-10 hospital managers who had a role in the implementation of nurse CPD. The interview explores hospitals' management, policies, barriers, and efforts in implementing nurse CPD. Interviews with hospital management were conducted simultaneously at almost the same time as the nurse's FGD.

   FGD on the Indonesian Nurses Association committee will be conducted on 8-10 committee members who have direct authority in the implementation of CPD. The FGD focuses on the policies, barriers, and efforts that professional organizations make on nurse CPD.

   The analysis and reflect stage or stage 3 of the 7 stages of this research will be carried out by analysing the results of the FGD. These results will used as a basis for determining strategic issues and potential solutions to the problems in this study.

   The interview will be conducted by 2 people, namely researchers and research assistants. Verbatim transcripts will be performed immediately after the interview is conducted by research assistants who follow the course of the interview.
2. Action

This stage will begin with the plan to change, the 4th stage of 7 stages of research. This stage aims to draw up an instructional design that will form the basis for the development of the e-CPD system. Activities will be carried out with a series of workshops 2 times to get mutual agreement. The workshop will be attended by nurse managers, The Indonesian Nurses Association representatives, clinical nurse assessors, and nurses in charge of care. The results of stage 4 will produce the Clinical Nurse II Competency Training Curriculum. At this stage, an expert review is also carried out to assess the suitability of the module preparation with existing provisions. Expert reviews will also be conducted to ensure that the curriculum has met the established rules. At this stage, researchers identify the ability of clinical nurses as the primary users, required features, learning media, assignments and assessments set.

The next stage is act, which is stage 5 of the 7 stages of research. This stage will carried out through the development of the e-CPD system. Researchers, in collaboration with IT professionals, will develop an e-CPD system designed to be able to facilitate the learning process as well as evaluation according to the curriculum that has been compiled. At this stage, the e-CPD system is also reviewed by the same experts who provide curriculum reviews. This is done so that the e-CPD system is built in accordance with the curriculum that has been prepared.

The observation stage, stage 6 of the 7 existing research stages, will carry out user testing. User testing aims to test the functionality of the e-CPD design that has been developed. User testing was carried out on 10 nurses who will become users of this system with the criteria: level I clinical nurses who work in hospitals, have gadgets and are willing to participate in the e-CPD system trial. The instruments used use the System Usability Scale (SUS). Participants will be asked to access and try all the features of the e-CPD application. Then, participants will be asked to complete an SUS questionnaire containing 10 questions through Google Forms. This questionnaire contains ease of access and possible use for these participants.

Reflect stage, is the last stage, stage 7 of the 7. At this stage, analysis and evaluation of the entire study that has been carried out and determine follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Level I clinical nurses who works in hospital
* Have a mobile device
* Willing to take e-CPD user testing

Exclusion Criteria:

* Did not complete the user testing

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
evaluating usability of e-CPD system, using System Usability Scale (SUS) instrumen, and Data will be collected using a Google form link given to participants after trying all the features in the e-CPD system. | Through study completion, an average of 3 months
  SUS has 10 questions and 5 answer choices. Answer choices range from strongly disagree to strongly agree. SUS has a minimum score of 0 and a maximum score of 100.
  After the calculation is carried out, the assessment results will be obtained. SUS assessment guidelines are as follow the acceptable score is approximately above 70 (above our average of 68), and the unacceptable score is below 50 (closely corresponding to our classification of scores below 51.6). They evaluated the range between 50 and 70 to be "marginally acceptable,"